CLINICAL TRIAL: NCT04506658
Title: Efficiency and Safety of High-frequency Radio Wave Electrotherapy With a Radio Frequency of 448 kHz in the Treatment of Patients With Organic Erectile Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Director for Research, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 07-20 from 15.04.2020
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Erectile Dysfunction
Keywords: high-frequency radio wave electrotherapy; radio frequency; 448 kHz
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: high-frequency radio wave electrotherapy with a frequency of 448 kHz on the penis structures.
- Control group (Sham Comparator)
  Interventions: Device: high-frequency radio wave electrotherapy with a frequency of 448 kHz on the penis structures.

INTERVENTIONS:
Device: high-frequency radio wave electrotherapy with a frequency of 448 kHz on the penis structures. — Patient in lithotomy position (supine) with return plate at lumbar level.
  Start with high power (within the allowed range) to get a faster hyperthermia and slowly decrease this percentage as the current builds up in the patient's body.
  Patients are undergoing high-frequency radio wave electrotherapy 2 times a week (12 procedures at all).
  Arms: Intervention group
Device: high-frequency radio wave electrotherapy with a frequency of 448 kHz on the penis structures. — Doctor uses sham sensor to reduce efficiency to zero.
  Arms: Control group

SUMMARY:
Efficiency and safety of high-frequency radio wave electrotherapy with a radio frequency of 448 kHz in the treatment of patients with organic erectile dysfunction. Sham comparator, parallel study including both the main and control group to demonstrate the efficiency of the device to treat erectile dysfunction.

DETAILED DESCRIPTION:
The objectives of this study are:

* To evaluate the effectiveness of the course treatment with the apparatus for continuous capacitive resistive monopolar electrotherapy with a radio frequency of 448 kHz in patients with organic erectile dysfunction.
* Assess the safety and tolerability of continuous capacitive resistive monopolar electrotherapy with a radio frequency of 448 kHz in patients with organic erectile dysfunction.
* To evaluate the duration of the effect of continuous capacitive resistive monopolar electrotherapy with a radio frequency of 448 kHz.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 79 years;
2. The diagnosis is confirmed by assessing the functional criteria of arterial factors of panel hemodynamics (dopplerography);
3. The diagnosis is confirmed by the assessment of the IIEF-5 questionnaire
4. Patients with organic erectile dysfunction lasting at least 6 months.
5. Patients with IIEF from 6 to 22 points.
6. Patients with a permanent sexual partner for more than 3 months;
7. Sexually Active Patients.

Non-inclusion criteria:

1. The use of other treatments for erectile dysfunction
2. Age under 18 and over 79 years old;
3. Anatomical deformation of the penis (angulation, cavernous fibrosis or Peyronie's disease);
4. The presence of diseases predisposing to the development of priapism (sickle cell anemia, multiple myeloma, leukemia, thrombocytopenia);
5. Running coagulation disorders;
6. The presence of tumors in the area of electrotherapy;
7. The presence of aneurysms in the propagation of radio frequency waves;
8. Angina pectoris;
9. Myocardial infarction, stroke, life-threatening arrhythmias;
10. Thrombosis, thromboembolic disease;
11. Arterial hypertension (blood pressure ≥ 170/90 mm Hg) or hypotension (blood pressure ≤ 90/50 mm Hg.);
12. The patient has a mental illness that does not allow an assessment of the effectiveness of therapy; history of alcoholism and drug addiction;

14. Active tuberculosis, chronic somatic diseases in the acute stage; 15. Condition after coronary artery bypass grafting (CABG); 16. Patient's involvement in another clinical trial in the last 3 months;

Exclusion Criteria:

1. Serious unwanted phenomenons associated with exposure to the apparatus.
2. Incorrect inclusion in the study.
3. A marked deterioration in the patient's condition due to an increase in the severity of the disease or the attachment of another disease.
4. The patient's appearance of non-inclusion criteria during the study.
5. Serious deviation from the protocol.
6. The desire of the patient or his legal representative.

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
A statistically significant increase in the number of points IIEF-5 | Through study completion, an average of 3 months after first procedure
  IIEF-5

SECONDARY OUTCOMES:
A statistically significant increase in penile blood flow. | Through study completion, an average of 3 months after first procedure
  According to Doppler
Statistically significant increase in SEP scores (Sexual Encounter Profile) | Through study completion, an average of 3 months after first procedure
  Schramek grading system score for assessing penile rigidity

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Korolev, M.D., Principal Investigator — Sechenov University
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.sechenov.ru
- See also: Related Info — http://www.urologypro.ru